CLINICAL TRIAL: NCT06609330
Title: Assessment and Treatment of Chronic Anger and Aggression Following Military-Related Interpersonal and Institutional Betrayal: A Pilot Investigation
Brief Title: Treatment of Chronic Anger and Aggression Following Military-Related Betrayal
Acronym: CART
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Principal Investigator, Vanessa Jacoby, Associate Professor, The University of Texas Health Science Center at San Antonio
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20230329HU; W81XWH-22-2-0085 (Other: United States Department of Defense)
Record Dates: First submitted 2024-08-14; First posted 2024-09-24 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Anger Problems; Aggression
Keywords: Anger management; Military-related betrayal; Deficit of trust
MeSH Terms: conditions — Aggression

STUDY DESIGN:
Intervention Model Description: Upon enrollment into the study, participants will begin with a minimal contact wait condition followed by randomization to different wait times (2-, 3-, or 4-weeks)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 2-week wait time group (Experimental): This group is randomized to a 2-week wait time prior to treatment with CART
  Interventions: Behavioral: Countering Chronic Anger and Aggression Related to Trauma and Transgressions (CART)
- 3-week wait time group (Experimental): This group is randomized to a 3-week wait time prior to treatment with CART
  Interventions: Behavioral: Countering Chronic Anger and Aggression Related to Trauma and Transgressions (CART)
- 4-week wait time group (Experimental): This group is randomized to a 4-week wait time prior to treatment with CART
  Interventions: Behavioral: Countering Chronic Anger and Aggression Related to Trauma and Transgressions (CART)

INTERVENTIONS:
Behavioral: Countering Chronic Anger and Aggression Related to Trauma and Transgressions (CART) — Countering Chronic Anger and Aggression Related to Trauma and Transgressions (CART), a novel intervention for reducing chronic anger and aggression and improving interpersonal relationships, in military personnel who have experienced military-related betrayal delivered in 14 treatment modules twice a week.
  Other Names: CART

SUMMARY:
The goal of this clinical trial is to learn if a treatment designed to deal with anger and aggression from a past betrayal will work. The study will be done on active duty military service members and veterans aged 18 or older. The main questions it aims to answer are:

* Will participants be satisfied with the treatment, and is the treatment feasible to do in a military outpatient setting
* Will the treatment help with anger and aggression issues.

Researchers will compare differences in groups that have different wait times (2-, 3-, or 4-weeks).

Participants will complete surveys before, during and after the treatment. The treatment will be 14 modules given twice a week. About 1 month after treatment ends, surveys will be taken again.

DETAILED DESCRIPTION:
Participants will undergo the study procedures described below. The preferred method of assessment and treatment is face-to-face in the STRONG STAR offices at Fort Cavazos. However, there may be circumstances when participants can complete the treatment through telebehavioral health (i.e., by phone or using a HIPAA-compliant video calling platform like Zoom). Decisions will be made on a case-by-case basis as issues arise for individuals (e.g., childcare) and in discussion with the treatment team. If participants do not have internet access they may need to complete assessments in person at the STRONG STAR office or by phone.

* During the wait time:

  * Complete a 5-10 minute assessment twice per week (Monday/Thursday or Tuesday/Friday) to assess level of anger, aggression, and interactions with others since last assessment.
  * The assigned therapist will call participants once a week for a 10-minute, check-in.
  * At the end of participants' assigned wait time, they will complete an assessment of level of anger, aggression, interactions with others, mental, and physical health.
* During treatment:

  * Begin treatment within 1 week of last wait time assessment.
  * Participate in 7-24 (average 14) one-hour bi-weekly (Monday/Thursday or Tuesday/Friday) CART sessions.
  * Prior to each session, participants will complete the same 5-10 minute assessment to assess level of anger, aggression, and interactions with others since last assessment.
  * At the final treatment session, participants will be scheduled to complete a 1-month follow-up assessment.
* For follow-up:

  * Complete a 1-month follow up assessment between 4-8 weeks after the final treatment session.
  * Participants will be sent a link to complete the follow-up assessment.
  * Complete the same questionnaires completed at pre-treatment plus an exit interview and a brief satisfaction survey.

ELIGIBILITY:
Inclusion Criteria:

* Adult active duty military service members and veterans aged 18 or older.
* Endorses a history of military-related betrayal (on the Modified Moral Injury Questionnaire)
* Endorses problematic anger in the past month (as evidenced by a score of 12 or above on the Dimensions of Anger Reactions; DAR-5)
* Engaged in at least 1 self-reported act of aggression in the past 1 month (on the Overt Aggression Scale-Modified; OAS-M)

Exclusion Criteria:

* Participated in an anger management or trauma-focused intervention within the past 3 months as assessed by self-report.
* Acute suicidality requiring immediate intervention, such as hospitalization as assessed by the Depressive Symptoms Index-Suicidality Subscale (DSI-SS) combined with follow up clinical interview for elevated scores.
* Is currently homicidal with plans and intent to hurt a specific person and requiring immediate intervention as measured by self-report and follow-up with clinician if screened positive.
* Moderate to severe brain injury as measured by inability to comprehend the informed consent document or baseline assessments.
* Has severe alcohol consumption patterns as evidenced by a score of 19 or above on the Alcohol Use Disorders Identification Test (AUDIT).
* Experiencing active psychosis or mania as measured by the Prodromal Questionnaire-Brief Version and the Mood Disorders Questionnaire.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Successful recruitment | Study start to last subject enrolled, approximately 1 year
  Number of eligible referrals that are recruited, enrolled into the study and randomized to treatment
Client satisfaction survey (CSQ-8) | 1 month after study end ( at approximately 11-18 weeks)
  The survey will assess participant acceptability using the CSQ-8, an 8-item self-report measure designed to assess client satisfaction. Each question is answered on a 4-point scale with a possible range of scores between 8-32. A higher score indicates a higher level of overall satisfaction. Mean scores will be used to determine participant satisfaction.
Overt Aggression Scale-Modified (OAS-M) | Baseline to 1 month post treatment (approximately 11-18 weeks)
  A 17-item measure that assesses frequency of different aggression acts in outpatient settings, including verbal and physical aggression against self, other, and objects. The OAS-M is scored by summing the instances of aggression since the last assessment. The OAS-M had been administered as an interview as well as self-report and will be administered as a self-report in this study, consistent with past aggression research with veterans (Miles, Kent et al., 2020). The score is calculated using a sum total of all instances of aggression. Higher scores indicate a greater frequency of aggressive behaviors.
Inventory of Interpersonal Problems-Short Version (IIP-32) | Baseline to 1 month post treatment (approximately 11-18 weeks)
  A 32-item self-report assessment designed to measure interpersonal functioning. Items are scored on a five-point scale from 0 (not at all) to 4 (extremely) in response to the stem: "How much have you been distressed by this problem?" There are 8 factors and a total score. The 8 factors are: hard to be assertive, hard to be sociable, hard to be supportive, too dependent, too caring, too aggressive, hard to be involved and too open. The possible total score ranges from a T-score are 0-100. T-scores that are higher than 60 are above average and T-scores 70 or higher suggest significant interpersonal difficulty.
State Trait Anger Expression Inventory-2 (STAXI-2) | Baseline to 1 month post treatment (approximately 11-18 weeks)
  A 57-item inventory which measures the frequency and intensity of anger as an emotional state. There are 6 scales, 5 subscales, and an Anger Expression Index (total anger expression). The State Anger scale (15 items) measures anger intensity as a momentary emotional state, while the Trait Anger scale (10 items) measures the disposition to experience angry feelings as a personality-like trait over lengthy time periods (i.e., the individual's disposition to become angry or angry temperament). The Anger Expression scale (16 items) and the Anger Control scale (16 items) measure four anger-related trait dimensions. Ratings of items are on a 4-point response scales that measure state anger (intensity) as well as trait anger (frequency). The possible total range is a T-score from 0 to 100. Individuals with anger scores higher than the 75-percentile experience and/ or express angry feelings to a degree that may interfere with optimal functioning.

SECONDARY OUTCOMES:
Rate of protocol completion | Treatment end (Approximately 7-14 weeks)
  The 14 modules may be completed within a 7-14 week time period by each participant.
Number of modules completed | Baseline to end of treatment (approximately 7-14 weeks)
  A count of how many of the 14 modules are completed
Brief Inventory of Psychosocial Functioning (B-IPF) | Baseline to 1 month post treatment (approximately 11-18 weeks)
  A 7-item, self-report measures of psychosocial functioning in seven life domains: romantic relationship, relationship with children, family relationships, friendships and socializing, work, training and education, and activities of daily living. In each area on a 7-point scale ranging from 0 = Not at all to 6 = Very much. The B-IPF total score is calculated by summing the scale items completed by the respondent, dividing by the maximum possible score based upon the number of applicable items and multiplying by 100. Higher scores indicate greater psychosocial dysfunction.
Dimensions of Anger Reactions (DAR-5) | Baseline to 1 month post treatment (approximately 11-18 weeks)
  A 5-item self report measure that assesses anger frequency, intensity, urge to act aggressively and impact on social functioning over the past 1 month. Respondents are asked how impacted they have been on a five-point Likert scale ranging from 0-5. Items are summed to provide a total severity score (range 5-25). A score of 12 or higher indicates problematic anger.
Revised Conflict Tactics Scale Short Form (CTS-2) | Baseline to 1 month post treatment (approximately 11-18 weeks)
  The CTS-2 poses 39 questions to assess five tactics used when conflict occurs within the relationships of dating, cohabitating, or marital couples. For this study, only the Physical Assault and Psychological Aggression subscales (20 items) of the CTS-2 will be used, broadening the assessment of conflict to query interpersonal conflict among friends, colleagues, and acquaintances as well as the family. The scoring range is: 0-6, Two Subscales: 1) Psychological Aggression: 1-8 2) Physical Assault: 9-20, Special Coding: Sum midpoints of chosen response option: Never-0, Once-1, Twice-2, 3-5 times -4 , 6-10 times-8, 11-20 times-15, greater than 20 times-25. For item scoring range 0-25, Psychological Aggression scoring range 0-200, Physical Assault scoring range 0-300. The higher scores indicate higher levels of Psychological Aggression and Physical Assault.
Trauma-Related Anger Scale (TRAS) | Baseline to 1 month post treatment (approximately 11-18 weeks)
  A 19-item self report measure to assess anger in the context of posttraumatic stress. Participants are asked to rate each item from Not at all true (0) to ;Definitely True(3) both prior to their traumatic event, and within the past two weeks. The scoring range for the items summed to provide a total severity score is 0-57. Items 1-7 = Anger giving a sense of control or energy, Items 8-14 = thought and emotional avoidance relating to anger, Items 15-17 = anger in response to threat, Items 18-19 = anger in response to pity. The higher score means greater anger in the context of PTSD. Higher scores in past two weeks, as compared with pre-trauma scores, indicate more severe trauma-related anger.

CONTACTS AND LOCATIONS:
Overall Officials: Vanessa Jacoby, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio; Alan Peterson, PhD, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Carl R. Darnall Army Medical Center (CRDAMC) at Fort Cavazos, Fort Cavazos, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
At the conclusion of the study all data will be stripped of identifiers. De-identified (anonymized) data will be maintained indefinitely in the STRONG STAR Repository. Identifiable data from participants who signed the consent to have their data placed in the STRONG STAR Repository will be maintained under the UTHSCSA IRB-approved Repository protocol indefinitely.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: At the conclusion of the study and after data are analyzed.
Access Criteria: Researchers who are interested in IPD should contact STRONG STAR at https://www.strongstar.org/contact/
URL: https://www.strongstar.org/contact/